CLINICAL TRIAL: NCT00377598
Title: A Phase 2, Double Blind, Placebo Controlled, Dose-Ranging Study in Subjects With Postherpetic Neuralgia (PHN) to Evaluate the Efficacy, Safety, Tolerability, and Pharmacokinetics of Four Doses of TAK-583, Compared With Placebo
Brief Title: Efficacy, Safety and Tolerability Study of TAK-583 in Subjects With Postherpetic Neuralgia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TAK-583-EC201; 2005-005863-26 (EudraCT Number); U1111-1127-6187 (Registry Identifier: WHO)
Record Dates: First submitted 2006-09-14; First posted 2006-09-18 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-01

CONDITIONS: Neuralgia, Postherpetic
Keywords: Herpes Zoster; Neuralgia; Drug Therapy
MeSH Terms: conditions — Neuralgia, Postherpetic; Herpes Zoster; Neuralgia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- TAK-583 5 mg QD (Experimental)
  Interventions: Drug: TAK-583
- TAK-583 25 mg QD (Experimental)
  Interventions: Drug: TAK-583
- TAK-583 50 mg QD (Experimental)
  Interventions: Drug: TAK-583
- TAK-583 100 mg QD (Experimental)
  Interventions: Drug: TAK-583
- Placebo QD (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TAK-583 — TAK-583 5 mg, tablets, orally, once daily for up to 8 weeks
  Arms: TAK-583 5 mg QD
Drug: TAK-583 — TAK-583 25 mg, tablets, orally, once daily for up to 8 weeks
  Arms: TAK-583 25 mg QD
Drug: TAK-583 — TAK-583 50 mg, tablets, orally, once daily for up to 8 weeks
  Arms: TAK-583 50 mg QD
Drug: TAK-583 — TAK-583 100 mg, tablets, orally, once daily for up to 8 weeks
  Arms: TAK-583 100 mg QD
Drug: Placebo — TAK-583 placebo-matching tablets, orally, once daily for up to 8 weeks
  Arms: Placebo QD

SUMMARY:
The purpose of this study is to evaluate the efficacy of TAK-583, once daily (QD), in relieving pain in subjects with postherpetic neuralgia.

DETAILED DESCRIPTION:
Postherpetic neuralgia is defined as neuropathic pain still present 3 months following healing of the herpes zoster rash. Symptoms of postherpetic neuralgia may include a complex combination of symptoms, including a deep aching, shooting or burning pain, sensory deficits, hyperalgesia, allodynia, paresthesia, and dysesthesia. Postherpetic neuralgia is more common in the elderly, and it can have a debilitating effect on a patient. The most commonly prescribed treatments are tricyclic antidepressants and anticonvulsants, however these treatments are effective in approximately half of subjects and may also have undesirable side effects (eg, dizziness and somnolence).

TAK-583 is a synthetic compound under development by Takeda Global Research & Development Center, Inc. as a treatment for neuropathic pain and for delaying the progression of diabetic neuropathy.

Individuals who want to participate in this study will be required to provide written informed consent. Study participation is anticipated to be about 11 Weeks. Multiple procedures will occur at each visit which may include fasting, blood collection, urine collection, vital signs, body height and weight, physical examinations and electrocardiograms.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects with postherpetic neuralgia whose pain has been present for >3 months following healing of the herpes zoster rash.
* Subjects with an mean pain intensity score of 4 or more (determined from at least 4 daily recordings of pain intensity on an 11-point numerical scale over the preceding 7 days) during the baseline phase.
* Subjects aged 50 years and above.
* The female subject is not of child-bearing potential (eg, sterilized, postmenopausal).

Exclusion Criteria:

* Malignancy within the past 2 years with the exception of basal cell carcinoma.
* Subjects who have undergone neurolytic or neurosurgical therapy for postherpetic neuralgia.
* Clinically significant, actively treated or unstable hepatic, biliary, respiratory, renal, rheumatologic, or hematologic illnesses, or unstable cardiovascular disease as assessed by the investigator.
* WBC less than 2500, ANC less than 1500, platelets less than 100,000; ALT, AST or alkaline phosphatase greater than 1.5x ULN; total bilirubin greater than or equal to 1.2 times the upper limit of normal (excluding Gilbert's Disease); predicted GFR using Cockcroft and Gault formula less than or equal to 40 mL/min.
* Subjects with greater than 5 red blood cells per high-power field on urinalysis.
* Subjects with an albumin/creatinine ratio in an untimed ("spot") morning urine specimen greater than the upper limit of normal.
* Subjects who are immunocompromised or have clinically significant haematological abnormalities.
* Subjects with a history of HIV infection.
* Subjects with a positive hepatitis panel (including hepatitis B surface antigen, antibody to hepatitis B core antigen, antibody to hepatitis B surface antigen, or antibody to hepatitis C virus), except subjects with positive antibodies to hepatitis B surface antigen who have received hepatitis B vaccination and who have no history of serological evidence of liver disease.
* Subjects having other severe pain which may impair the self assessment of the pain due to postherpetic neuralgia.
* Subjects who have participated in a clinical trial for an investigational drug and/or agent within 30 days prior to baseline.
* Subjects who have received TAK-583 in a previous clinical study.
* Subjects who have donated more than 400 mL of blood in the 90 days prior to the beginning of the study.
* Subjects who have a history of alcohol or illicit drug abuse in the past 2 years
* Clinically significant abnormal 12 lead electrocardiogram, including QT interval corrected for heart rate greater than 450 ms that is confirmed on a repeat electrocardiogram.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 399 (Actual)
Dates: Start 2006-10; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in average daily pain intensity score for the previous 7 days | Week 8 or Final Visit

SECONDARY OUTCOMES:
Change from baseline to each study visit in average daily pain intensity score for the last 7 days | At All Visits
Change from baseline in pain assessment as assessed by Short form McGill Pain Questionnaire | Week 8 or Final Visit
Change from baseline in weekly mean sleep interference scores (assessed on an 11-point numerical scale in the subject's sleep diary) | Week 8 or Final Visit
Clinician and subject global impression of change using a 7-point scale | Week 8 or Final Visit
Change from baseline in quality of life as assessed by Short Form-36 | Week 8 or Final Visit
Change from baseline in Profile of Mood States | Week 8 or Final Visit
Proportions of subjects with at least 30% and 50% reduction from baseline in average daily pain intensity score | Week 8 or Final Visit

CONTACTS AND LOCATIONS:
Overall Officials: VP Clinical Science, Study Director — Takeda Global Research & Development Center
Locations (48):
- Australia (7):
  - Sydney, New South Wales
  - Kipparing, Queensland
  - Maroochydore, Queensland
  - Box Hill, Victoria
  - Carlton, Victoria
  - Fitzroy, Victoria
  - Perth, Western Australia
- Sofia, Bulgaria
- Czechia (5):
  - Hradec Králové
  - Moravská Ostrava
  - Olomouc
  - Ostrava
  - Pilsen
- Germany (9):
  - Berlin
  - Dresden
  - Frankfurt
  - Görlitz
  - Hamburg
  - Jena
  - Leipzig
  - Magdeburg
  - Schwerin
- Netherlands (6):
  - Arnhem
  - Breda
  - Roosendaal
  - Rotterdam
  - Stadskanaal
  - Utrecht
- Poland (4):
  - Gdansk
  - Lublin
  - Mosina k/Poznania
  - Poznan
- Russia (3):
  - Kazan'
  - Moscow
  - Saint Petersburg
- South Africa (8):
  - Bloemfontein, Free State
  - Pretoria, Gauteng
  - Amanzimtori, KwaZulu-Natal
  - Durban, KwaZulu-Natal
  - Breyten, Mpumalanga
  - Mbombela, Mpumalanga
  - Polokwane, Western Cape
  - Worcester, Western Cape
- United Kingdom (5):
  - Chichester
  - Darlington
  - Glasgow
  - Plymouth
  - Solihull